CLINICAL TRIAL: NCT03383627
Title: Assessment of Glycemic Control in Patients With Type 2 Diabetes Mellitus and Late Stage Chronic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Lubaina Presswala, Principal Investigator, Northwell Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 17-0531
Record Dates: First submitted 2017-10-30; First posted 2017-12-26 (Actual); Results first posted 2020-04-07 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-03

CONDITIONS: Diabetes; Kidney Diseases
Keywords: Chronic Kidney Disease
MeSH Terms: conditions — Diabetes Mellitus; Kidney Diseases; Renal Insufficiency, Chronic | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Continuous glucose monitoring (Experimental): * If subjects meet inclusion criteria then they will return to the research site on Day 1 to place Freestyle Libre Pro device by the research staff for 14-day monitoring.
  * Subjects will be advised to return to the research site on Day 14 to remove the CGM device for analysis. On Day 14, blood will be drawn for HbA1c and fructosamine, The blood drawn for this research will be approximately 10-15 milliliters.
  * There are no drug washout periods. Subjects will continue to take all their medications and/or insulins as prescribed by their doctor.
  * Baseline data including age, race, ethnicity, past medical history, home medication list, and diabetes related laboratory data will be collected.
  Interventions: Device: Continuous Glucose Monitoring

INTERVENTIONS:
Device: Continuous Glucose Monitoring — * The FreeStyle Libre Pro Flash Glucose Monitoring System is a professional continuous glucose monitoring (CGM) device indicated for detecting trends and tracking patterns in persons (age 18 and older) with diabetes. The Freestyle Libre Pro device is FDA approved (PMA# P150021). Participants will use the FreeStyle Libre Pro Flash Glucose Monitoring device according to its approved use, on the back of the arm.
  * CGM monitoring will be performed on Day 1 by placing the Freestyle Libre Pro on research subjects for intended use of 14 days.
  * Subjects will be advised to return to the research site on Day 14 to remove the CGM device for analysis.

SUMMARY:
Diabetes control is often assessed by tests of glucose levels over time, such as the glycosylated hemoglobin A1c (HbA1c) and fructosamine. In the later stages of chronic kidney disease (CKD) there is limited data available on the utility of these tests. There are reasons to believe that the tests may be less accurate in this population. Continuous glucose monitoring (CGM) offers an effective method for understanding the totality of glucose exposure and incidence of both hyperglycemic and hypoglycemic excursions.

DETAILED DESCRIPTION:
In the proposed study Investigator plan to utilize CGM in patients with late stage CKD stages 3b-5 to 1) determine accuracy of HbA1c and serum fructosamine testing as measures of glucose control in patients with Type 2 Diabetes Mellitus (T2DM), 2) Better understand test characteristics in the late stage CKD population (correlation, linear equation, slope, Y intercept, average glucose at different HbA1c levels), 3) Develop a preliminary understanding of how test characteristics differ in late stage CKD compared to other patients with diabetes, 4) quantify time burden and number of episodes of hypoglycemia, 4) study hyperglycemic burden and 5) analyze glucose variability. The research staff will explain the study to patients that meet all inclusion criteria. Patients will get time to understand the study, review the consent document, ask questions to the PI, and then provide their consent to participate in the study. On Day 1 of the study, a CGM (Freestyle Libre) device will be placed on patients with CKD 3b-5 which will be worn for 14 consecutive days. Patients will return on Day 14 to remove the CGM device. HbA1c and fructosamine values will be drawn on Day 14 and these results will be compared with average glucose monitoring values as recorded on the CGM device. Incidence, duration, and severity of both hypoglycemic and hyperglycemic events will be analyzed. Investigators hypothesis that there will be significant variability in the serum HbA1c values when compared with calculated HbA1c from CGM readings. Investigators also hypothesize that the results will reflect a greater incidence of hypoglycemia in this population by CGM analysis.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older with ability to speak and understand English
* Established diagnosis of type 2 Diabetes Mellitus
* Chronic Kidney Disease (stages 3b, 4 or 5, eGFR (Glomerular Filtration Rate) < 45 ml/min, and not on dialysis) documented within 3 months of enrollment

Exclusion Criteria:

* Type 2 Diabetes Mellitus.
* Patient with End stage kidney disease on Dialysis.
* Presence of Hemoglobinopathies.
* Red blood cell transfusion in the last 12 weeks.
* Hb < 9 g/dL documented within 3 months of enrollment - Dosing with an erythropoiesis stimulating agent is acceptable but dose must be stable for two months.
* Use of acetaminophen on a daily basis.
* Systemic steroid treatment in the past 12 weeks.
* Greater than 50% dose change in diabetes medications or new diabetes medications started in the previous 8 weeks.
* Currently pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2018-08-21 (Actual); Study Completion 2018-08-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lubaina Presswala, DO, Principal Investigator — Northwell Health
Locations (1):
- Northwell Health (Division Endocrinology and Nephrology), Great Neck, New York, United States

IPD SHARING:
Plan to Share IPD: No
Access to study data will be limited to Institutional Review Board (IRB) approved personnel only.

REFERENCES:
- [Background] Miedema K. Standardization of HbA1c and Optimal Range of Monitoring. Scand J Clin Lab Invest Suppl. 2005;240:61-72. doi: 10.1080/00365510500236143. PMID 16112961
- [Background] Rabkin R, Ryan MP, Duckworth WC. The renal metabolism of insulin. Diabetologia. 1984 Sep;27(3):351-7. doi: 10.1007/BF00304849. PMID 6389240
- [Background] Castellino P, DeFronzo RA. Glucose metabolism and the kidney. Semin Nephrol. 1990 Sep;10(5):458-63. PMID 2236987
- [Background] Dolscheid-Pommerich RC, Kirchner S, Weigel C, Eichhorn L, Conrad R, Stoffel-Wagner B, Zur B. Impact of carbamylation on three different methods, HPLC, capillary electrophoresis and TINIA of measuring HbA1c levels in patients with kidney disease. Diabetes Res Clin Pract. 2015 Apr;108(1):15-22. doi: 10.1016/j.diabres.2015.01.034. Epub 2015 Jan 29. PMID 25684605

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Continuous Glucose Monitoring
Started | 80
Completed | 80
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Continuous Glucose Monitoring
Number analyzed (Participants) | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.3 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 61
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 77
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 11
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 53
  More than one race | 1
  Unknown or Not Reported | 4
Cause of Chronic Kidney Disease [Count of Participants; unit: Participants]
  Diabetes Mellitus Type 2 | 63
  Others | 17
Medical History [Count of Participants; unit: Participants]
  Congestive Heart Failure | 20
  Coronary Artery Disease | 26
  Hypertension | 77
  History of Stroke | 17
  History of Maliganancy | 6
eGFR [Count of Participants; unit: Participants]
  0 to <=15 mL/min | 15
  >15 to <=30 mL/min | 34
  >30 to <=45 mL/min | 31
BMI [Count of Participants; unit: Participants]
  <=25 | 14
  >25 to <=30 | 33
  >30 to >=35 | 21
  >35 | 12

OUTCOME MEASURES:

1. Primary Outcome: Mean Glucose Concentration Measured by CGM
Description: Mean glucose concentration (mg/dL) will be measured using measurements taken by CGM device.
Time Frame: 14 Days
Measure: Mean (Inter-Quartile Range); unit: mg/dL
Groups:
- Continuous Glucose Monitoring: Subjects enrolled and wearing CGM device
Arm/Group | Continuous Glucose Monitoring
Number analyzed (Participants) | 80
mg/dL | 151.5 [75 to 405]

2. Primary Outcome: Number of Participants With Hypoglycemic Events
Description: Hypoglycemic event will be considered when blood sugar level is <=70 mg/dl. Detail information like time of event, number of subjects with an event, duration of event will be analyzed.
Time Frame: 14 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Continuous Glucose Monitoring
Number analyzed (Participants) | 80
Participants | 61

3. Primary Outcome: Mean Number of Hypoglycemic Events Per Participant.
Description: Total number of hypoglycemic events per subject will be calculated during the study period. Mean number of events per subject will be analyzed.
Time Frame: 14 Days
Measure: Mean (Standard Deviation); unit: Hypoglycemic events
Arm/Group | Continuous Glucose Monitoring
Number analyzed (Participants) | 80
Hypoglycemic events | 7.5 (9.0)

4. Primary Outcome: Duration Hypoglycemic Events
Description: As monitoring device measures blood glucose level numerous time, duration of hypoglycemic event will be calculated in percent time per subject based on total duration of time subject wore CGM device.
Time Frame: 14 Days
Measure: Mean (Standard Deviation); unit: Percentage time with Hypoglycemia
Arm/Group | Continuous Glucose Monitoring
Number analyzed (Participants) | 80
Percentage time with Hypoglycemia | 7.5 (10.1)

5. Primary Outcome: Mean HbA1c
Description: HbA1c collected at end of the participation.
Time Frame: 14 Days
Measure: Mean (Inter-Quartile Range); unit: mmol/mol
Arm/Group | Continuous Glucose Monitoring
Number analyzed (Participants) | 80
mmol/mol | 7.2 [4.8 to 13.2]

6. Secondary Outcome: Mean Serum Fructosamine Concentration
Description: Serum fructosamine (µmol/L) collected at the end of participation.
Time Frame: 14 Days
Measure: Mean (Inter-Quartile Range); unit: µmol/L
Arm/Group | Continuous Glucose Monitoring
Number analyzed (Participants) | 80
µmol/L | 304.1 [177 to 523]

7. Secondary Outcome: Determination of Serum Fructosamine
Description: Using blood glucose information measured with continuous blood glucose monitoring device, probable level of serum fructosamine (µmol/L) will be measured for each participant and mean will be analyzed.
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Continuous Glucose Monitoring
Number analyzed (Participants) | 80
µmol/L | 304.1 (57.2)

ADVERSE EVENTS:
Time Frame: Over the period of study participation (Up to 14 days from date of enrollment).
Arm/Group | Continuous Glucose Monitoring
All-Cause Mortality (participants affected / at risk) | 0/80
Serious Adverse Events (participants affected / at risk) | 0/80
Other Adverse Events (participants affected / at risk) | 0/80

LIMITATIONS AND CAVEATS:
The sample size of 80 patients were predominately male and non-Hispanic. It would also have been meaningful to have more robust data of a diary of self-reported symptoms during the 14 day period.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-06-22): https://cdn.clinicaltrials.gov/large-docs/27/NCT03383627/Prot_SAP_000.pdf
  • Informed Consent Form (2018-06-22): https://cdn.clinicaltrials.gov/large-docs/27/NCT03383627/ICF_001.pdf